CLINICAL TRIAL: NCT02272452
Title: Assistance in Neurosurgery by Extemporaneous Analysis of Magnetic Resonance of the Metabolic Content in Excised Tissues (ExtempoRMN)
Brief Title: Assistance in Neurosurgery (ExtempoRMN)
Acronym: ExtempoRMN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: ExtempoRMN - RNI
Record Dates: First submitted 2014-10-15; First posted 2014-10-23 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Primary Brain Tumor; Glioma
Keywords: High resolution magic angle spinning Nuclear magnetic resonance; Nuclear magnetic resonance; Spectroscopy; Primary brain tumors; Gliomas; extemporaneous analysis
MeSH Terms: conditions — Brain Neoplasms; Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: High-Resolution Magic-Angle Spinning Nuclear Magnetic Resonance spectroscopy
  Other Names: HRMAS-NMR

SUMMARY:
The main ambition of this project is to develop, and provide the medical community, an innovative method to analyze extemporaneously, during a neurosurgery operation, excised tissues. This method is based on the analysis of the metabolic profile of excised tissues by the technique of High-Resolution Magic-Angle Spinning (HR-MAS) Nuclear Magnetic Resonance (NMR) spectroscopy. Indeed HRMAS NMR method can provide in a sufficiently short time lapse (currently about 30 minutes but within our project a time lapse of 15 min or even less is ultimately intended), medical information that can complement those obtained by classic histological examination.

Primary purpose:

The main objective of this study is to determine the sensitivity of HRMAS NMR spectroscopy in detecting residual tumor infiltration at the brain resection cavity. The investigators aim to determine the relevance of the metabolic analysis compared to histological analysis during a neurosurgery operation. This involves analyzing excised tissue samples, obtained from the operating rooms of Strasbourg University Hospitals, and Colmar Hospital Center, with no return to neurosurgeon for surgery.

Secondary purposes:

The secondary objectives of the protocol are to investigate the metabolome of different types of brain tumors, in order to find prognostic and diagnostic markers. It consists in detecting metabolomic factors of bad prognosis, and potential marker of good prognosis such as the IDH mutation.

ELIGIBILITY:
Inclusion criteria:

* Male or female
* Age 18 years of age or older at the time of surgery
* Primary brain tumors (gliomas mainly) or epilepsy, for which neurosurgical intervention is programmed
* In the case of brain tumors: primary-lesions or transformation of low-grade gliomas into high-grade gliomas not treated with radiotherapy
* Affiliated with a social security
* Having signed the informed consent
* Having been informed of the results of the medical examination prior

Exclusion criteria:

* Relapse of tumors previously treated with radiotherapy or chemotherapy
* Subject under treatment (radiotherapy or chemotherapy) prior to surgery
* Metastatic lesions (location of the primary lesion outside the central nervous system)
* Inability to give to the subject or his/her family enlightened information (subject in emergency situation, difficulties of understanding...)
* Subject under judicial protection
* Subject under guardianship or curatorship
* Patients' Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Under the " ExtempoRMN "project, we propose to focus on primary brain tumors mainly gliomas that include: Glioblastomas, the low-grade oligodendrogliomas (WHO grade II) and high grade (WHO grade III), Astrocytomas. Normality will be obtained by analysis of control brain tissues from epilepsy surgery. Study population for this project is all the patients of department of neurosurgery of Strasbourg University Hospitals and Colmar Hospital center, for whom a neurosurgical operation is programmed before inclusion in this study, and who meets inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The percentage of the cases for which, the HRMAS NMR spectroscopy results of the excised tissues are consistent with quantitative histological analysis of the same excised tissues. | 3 years from the beginning of the study
  To validate the primary endpoint of this study, statistical analysis should confirm this consistency in at least 95% of the cases.

CONTACTS AND LOCATIONS:
Overall Officials: Izzie Jacques Namer, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (3):
- France (3):
  - Service de Biophysique et de Médecine Nucléaire, Hôpital de Hautepierre, Strasbourg
  - Service de neurochirurgie, Strasbourg
  - Service de Neurochirurgie, Strasbourg